CLINICAL TRIAL: NCT01108380
Title: Evaluation of Liver Regeneration With Autologous Peripheral Stem Cells Transplantation in the Patient Needed Extensive Hepatectomy
Brief Title: Evaluation of Liver Regeneration With Autologous Peripheral Stem Cells
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other)
Responsible Party: Ho-Seong Han. Chairman of surgery department. Seoul National University Bundang Hospital, Surgery department
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNUBH-GS-HBP3; B-0901-068-003 (Other: Seoul National University Bundang Hospital)
Record Dates: First submitted 2010-04-20; First posted 2010-04-22 (Estimated); Last update posted 2010-12-15 (Estimated); Status verified 2010-12

CONDITIONS: Liver Cirrhosis
Keywords: Liver cirrhosis; liver regeneration; liver volume; liver function; hepatocellular carcinoma, extensive; hepatectomy
MeSH Terms: conditions — Liver Cirrhosis; Carcinoma, Hepatocellular | interventions — Plasmapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1. CD34 (Experimental): 1. 4 days injection of G-CSF (10μg/kg, Subcutaneous infusion)
  2. On 5th day, plasmapheresis will be performed to select mononuclear cells. (at least 4x10(9) of mononuclear cells)
  3. CD 34 cells will be selected by CliniMACS (Miltenyi Biotec, Bergisch- Gladbach, Germany) (at least 1x10(7) of CD 34 cell)
  4. In same day, right portal vein embolization with infusion of CD 34 cells into left portal vein will be performed.
  Interventions: Procedure: Plasma pheresis, Right portal vein embolization
- 2. Mononucelar cell (Active Comparator): 1. 4 days injection of G-CSF (10μg/kg, Subcutaneous infusion)
  2. On 5th day, plasma pheresis will be performed to select mononuclear cells. (at least 4x10(9) of mononuclear cells)
  3. In same day, right portal vein embolization with infusion of mononuclear cells into left portal vein will be performed.
  Interventions: Procedure: Plasma pheresis, Right portal vein embolization
- 3. Control (Other): Without infusion of G-CSF, patients will be performed just right portal vein embolization
  Interventions: Procedure: Plasma pheresis, Right portal vein embolization

INTERVENTIONS:
Procedure: Plasma pheresis, Right portal vein embolization — Plasma pheresis : With insertin of 2 intravenous line, plasmapheresis will be done with COBE BCT Inc. It will be performed under supervision of clinical laboratorians and doctors.
  Right portal vein : Under ultrasonography guided, left portal vein be punctured. Right portal vein will be embolized by coil or gelfoam.
  Other Names: COBE BCT Inc : for plasmapheresis

SUMMARY:
For patient with liver cirrhosis who need to right or extended right hepatectomy, we will treat with autologous peripheral stem cells transplantation to facilitate liver regeneration. We will asses liver regeneration by evaluation of liver volume and liver function test.

DETAILED DESCRIPTION:
1. Patients: 30 patients (10 patients in each 3 group)
2. Indication:

   * Patients with Primary hepatocellular carcinoma combined liver cirrhosis (Hepatitis B, C, Non-B Non-C)
   * Planned to right hepatectomy or extended right hepatectomy
   * Patients who need right portal vein embolization due to insufficient expected remnant liver volume (< 40%) or severe hepatic dysfunction(ICGR15>10%)
   * Child A classification
   * ICG R15 < 25%
   * Age : 20 - 70 years old
   * Expected life period > 3months
   * The patients who agreed to this study.
3. Contraindication

   * Patients who planned liver transplantation
   * Age <20 or >70 years old
   * Pregnant women
   * Patients on acute infection
   * Acute hepatic failure
   * Child class B or C
   * Heart failure
   * Existence of bleeding tendency : platelet < 30,000, INR > 2.2, Cr >2.5
   * Patients who did not agree to this study.
4. Allocation: We will allocate patients randomly to three group including control group.
5. Methods

   * Group 1: 4 days injection of G-CSF -> Plasma pheresis, Selection of CD34 cell -> Right portal vein embolization and infusion of CD34 cell into left portal vein.
   * Group 2: 4 days injection of G-CSF -> Plasma pheresis -> Right portal vein embolization and infusion of mononuclear cell into left portal vein.
   * Group 3 (control): Right portal vein embolization

   ( -> after 4 weeks, operation will be performed)
6. Evaluation: Change of liver volume, liver function test before and after portal vein embolization

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Primary hepatocellular carcinoma combined liver cirrhosis (Hepatitis B, C, Non-B Non-C)
2. Planned to right hepatectomy or extended right hepatectomy
3. Patients who need right portal vein embolization due to unsufficient expected remnant liver volume (< 40%) or severe hepatic dysfunction (ICG R15 > 10%)
4. Child A classification
5. ICG R15 < 25%
6. Age: 20 - 70 years old
7. Expected life period > 3months
8. The patients who agreed to this study

Exclusion Criteria:

1. Patients who planned liver transplantation
2. Age < 20 or > 70 years old
3. Pregnant women
4. Patients on acute infection
5. Acute hepatic failure
6. Child class B or C
7. Heart failure
8. Existence of bleeding tendency : platelet < 30,000, INR > 2.2, Cr >2.5
9. Patients who did not agree to this study

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Safety and efficacy, short term outcome | 4 weeks after procedure
  After portal vein embolization, we will compare liver volume by CT and liver function test by blood test in 3 groups. (Second and forth week)

SECONDARY OUTCOMES:
Safety and efficacy. | 12 weeks
  After 4 weeks of portal vein embolization, hepatectomy woul be performed in indicated patients. After hepatectomy, until 12 weeks, we will compare remnant liver volume by CT and liver function test by blood test.

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Seong Han, PhD, Principal Investigator — Chairman of surgery, Seoul National University Bundang Hospital
Locations (1):
- Ho-Seong Han, Seongnam-si, Gyeonggi-do, South Korea